CLINICAL TRIAL: NCT04594317
Title: Effect of Low Level Laser Therapy (LLLT) Versus Calcium Hydroxide Intra-canal Medication on Postoperative Pain and Total Amount of Substance P and IL-8 in Periapical Fluids in Patients With Symptomatic Apical Periodontitis: a Randomized Clinical Trial
Brief Title: Effect of Low-level Laser Therapy Versus Calcium Hydroxide Intracanal Medication on Postoperative Pain and Substance P Levels in Patients With Symptomatic Apical Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Radhwa Refaat Otaify, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENDO 3/3/5
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain; Apical Periodontitis
Keywords: low level laser therapy; calcium hydroxide; postoperative pain; biomarker; substance P; interleukin 8
MeSH Terms: conditions — Pain, Postoperative; Periapical Periodontitis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: randomized parallel clinical trial
Who Masked: Participant
Masking Description: The participants will be blinded to the study hypothesis as to which intervention is expected to be better.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low level laser therapy (Experimental): 970 ± 15-nm diode laser (Biolase Epic X, Biolase, Irvine, California, USA)will be activated at 0.5 W and 10 Hz at a distance of approximately 10 mm to the tissue around the apex of the root. A circular movement will be performed during application. Pulse duration will be 0.5 s, and pulse pause will be 50%. Total application time will be30 s for the tooth. For this application, a 200-μm optical tip will be used.
  Interventions: Device: low level laser therapy
- Calcium hydroxide intracanal medication (Active Comparator): calcium hydroxide paste (Metapaste, Meta Biomed Co., Ltd, Korea) will be inserted in the canal using disposable plastic tip and placed at a distance 1 or 2 mm less than the working length.
  Interventions: Device: low level laser therapy

INTERVENTIONS:
Device: low level laser therapy — buccal application of diode laser on non-contact mode

SUMMARY:
a randomized clinical study to compare the effect of using low level laser therapy versus calcium hydroxide intra-canal medication on:

* Incidence and intensity of postoperative pain in patients with symptomatic apical periodontitis.
* The intensity of postoperative percussion pain in patients with symptomatic apical periodontitis
* The total amount of substance P and Interleukin 8 in periapical fluids one week post instrumentation.

DETAILED DESCRIPTION:
Diagnosis:

Personal data including name, address and phone number in addition to medical history (Appendix II) and dental history (Appendix III) will be collected by the operator from each patient in specific forms, then history of chief complaint will be recorded. The selected patients should show symptoms of irreversible pulpitis. The operator will perform extra-oral and intra-oral clinical examination as the expected tooth to be included in this study should be examined tentatively using a diagnostic mirror and probe. Radiograph will be taken using bisecting angle technique with a periapical digital sensor plate1. The radiograph will help to identify if there is widening of periodontal ligament space, periapical radiolucency, deep caries near the pulp chamber or recurrent caries under restoration.

The diagnosis of symptomatic apical periodontitis is confirmed through:

* The patient history of pain with biting and confirmed with positive percussion test.
* After completing the diagnosis (symptomatic apical periodontitis) and confirming that the patient fulfills the eligibility criteria, the patient will be enrolled in the study. The treatment will be done in two visits.

Treatment procedure:

After diagnosing the case as symptomatic apical periodontitis and confirming that the patient conforms to all eligibility criteria, patients will be enrolled in in the study. Preoperative percussion pain level will be recorded using modified VAS. Treatment of all cases will be completed in two visits.

1. Anesthetizing the tooth using infiltration technique by local anesthesia of 1.8 ml of 4% Articiane with 1:100,000 epinephrine (Artinibsa®; Inibsa Dental, Lliçà de Vall,Spain)
2. Caries and/or coronal restorations will be removed completely with sterile bur and rubber dam will be applied.
3. Operative field, including the tooth, the clamp, and rubber dam sheet will be cleaned with 30% hydrogen peroxide until no further bubbling of the peroxide occurred. All surfaces will then be disinfected by a sterile cotton swab with a 5.25% sodium hypochlorite solution.
4. Access cavity will be prepared using another sterile round carbide bur size 3 and Endo-z bur(Dentsply Maillefer, Ballaigues, Switzerland)
5. After completing the access, the operative field and the pulp chamber will be cleaned and disinfected once again in the same way mentioned above. NaOCl will be then neutralized with 5% sodium thiosulfate.
6. Patency of the root canal will be confirmed using stainless steel handK-files size

   #10 and #15(K-Files, MANI, INC., Industrial Park, Utsunomiya, Tochigi, Japan).Working length will be determined using an electronic apex locator(Root ZX, J. Morita USA, Irvine, CA)then confirmed radiographically to be 1 mm shorter than radiographic apex. Then the canal will be enlarged to size #20.
7. Mechanical preparation will be done using M PRO rotary files in an endodontic motor(X-Smart, Dentsply Maillefer, USA). The first file (18/.09) will be used as an orifice opener for two thirds of the working length followed by (20/.04) and (25/.06) for the full working length and finally (35/.06). In-and-out motions will be applied with stroke lengths not exceeding 3 mm in the cervical, middle, and apical thirds until attaining the established WL. The first file is used with a continuous rotary motion at a speed of 500rpm and torque of 3Ncm. The second, third and fourth files are used with a speed of 300 rpm and torque of 1.5Ncm. The canal will be irrigated and recapitulated after the use of each instrument.
8. The canal will be thoroughly irrigated with 2.5% sodium hypochlorite root canal irrigant (5ml for 1 min) using disposable plastic syringe with side vented needle gauge 30 (Steri irrigation tips; Diadent, Chungcheongbuk-do, Korea) reaching 1 mm short of the working length. All teeth will receive the same volume of irrigant (5 ml prior to instrumentation, 5 ml between each file and 5 ml as final flush after root canal instrumentation to reach a total volume of 25 ml in total).
9. The canal will then be dried by using sterile paper points(Meta Biomed Co., Ltd, Korea) and then flushed with 5 ml of saline to inactivate the NaOCl. The postinstrumentation periapical sample (PS-1) will be collected after cleaning and shaping by introducing a fine sterile size 20 paper point 2 mm beyond the canal terminus for 1 min.This procedure will be performed twice. The paper points will be placed in a sterile micro-centrifugation tube (Merck) containing 2 mL of sterile physiological saline solution, and immediately transferred to a -80 °C freezer until further processing.
10. The patients will then be assigned into two groups (n = 23), as follows:

    * LLLT Group: 970 ± 15-nm diode laser (Biolase Epic X, Biolase, Irvine, California, USA)will be activated at 0.5 W and 10 Hz at a distance of approximately 10 mm to the tissue around the apex of the root. A circular movement will be performed during the application. Pulse duration will be 0.5 s, and pulse pause will be 50%. Total application time will be30 s for the tooth. For this application, a 200-μm optical tip will be used.
    * Calcium hydroxide Group: calcium hydroxide paste (Metapaste, Meta Biomed Co., Ltd, Korea) will be inserted in the canal using disposable plastic tip and placed at a distance 1 or 2 mm less than the working length.
11. The access cavity will be closed using sterile cotton pellet and temporary filling and patients will be recalled after 1 week.
12. The patients will record the incidence of pain and the pain level on modified VAS scale at 6,12, 24 and48 hours
13. In the recall appointment after 1 week. Rubber dam will be applied and tooth will be disinfected as before. The previously sampled canal will be re-entered, flushed with copious saline irrigation and a second periapical sample (PS-2) will be taken. After the sampling, final flush with 2.5% NaOCL and 17% EDTA will be done in both groups. Master cones of (0.40) taper gutta-percha(Meta Biomed Co., Ltd, Korea) will be fitted to the working length and a radiograph will be taken to ensure proper length. Obturation will be done by modified single cone technique using epoxy resin sealer(Adseal, Meta Biomed CO.,LTD, Korea)and 4% taper gutta percha cones together with auxillary cones.
14. The access cavity will be restored with composite resin and occlusal contact will be checked. The details of the endodontic procedure for each patient will be recorded in the patient's procedure chart

ELIGIBILITY:
Inclusion Criteria:

* Patients who are free from any physical or mental handicapping condition with no underlying systemic disease.
* Age between 25-50 years old.
* Males & Females.
* Single canaled teeth:

  * Diagnosed clinically with symptomatic apical periodontitis.
  * Widening in the periodontal membrane space or with small sized periapical radiolucency
  * Presence of pain with percussion and preoperative percussion pain level will be evaluated and recorded using modified visual analog scale (VAS).
* Patients' acceptance to participate in the trial.
* Patients who can understand pain scale and can sign the informed consent

Exclusion Criteria:

* Medically compromised patients: Pain levels and healing following treatment would be compromised as these patients have shown higher incidence of pain and lower healing rate.
* Pregnant women: Avoid radiation exposure, anesthesia, and medication.
* If analgesics or antibiotics have been administrated by the patient during the past 24 hours preoperatively might alter their pain perception.
* Patients reporting bruxism or clenching: Avoid further pressure on an already inflamed tooth inducing subsequent irritation and inflammation.
* Teeth that shows association with acute periapical abscess and swelling: Need special treatment steps which could involve additional visits with incision and drainage. Also, it could influence initiation and progression of postoperative pain.
* Greater than grade I mobility or pocket depth greater than 5mm. Need special surgical and/or periodontal therapy.
* No restorability: Hopeless tooth.
* Immature teeth.
* Radiographic evidence of external or internal root resorption vertical root fracture, perforation, calcification.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative pain | 24 hours
  incidence of postoperative pain will be recorded in pain chart

SECONDARY OUTCOMES:
intensity of postoperative pain: modified visual analogue scale | 48 hours
  intensity of postoperative pain will be recorded using modified visual analogue scale ( it's a scale from 0-10 , in which 0 represents lowest pain level with NO pain and 10 represents the highest pain level).

IPD SHARING:
Plan to Share IPD: Undecided
Still to decide whether to share it or not